CLINICAL TRIAL: NCT03263572
Title: Phase II Study of the Combination of Blinatumomab and Ponatinib in Patients With Philadelphia Chromosome (Ph)-Positive and/or BCR-ABL Positive Acute Lymphoblastic Leukemia (ALL)
Brief Title: Blinatumomab, Methotrexate, Cytarabine, and Ponatinib in Treating Patients With Philadelphia Chromosome-Positive, or BCR-ABL Positive, or Relapsed/Refractory, Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Amgen (Industry); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0792; NCI-2018-01078 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0792 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Lymphoblastic Leukemia; BCR-ABL1 Fusion Protein Expression; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Philadelphia Chromosome Positive; Recurrent Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia; t(9;22)
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis | interventions — blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Cytarabine; Methotrexate; merphos; ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (blinatumomab, chemotherapy, ponatinib) (Experimental): Patients receive blinatumomab IV nonstop on days 1-28 of cycles 1-5, and methotrexate and cytarabine intrathecally (by spinal tap) on days 1, 15, and 29 of cycles 1-4. Patients also receive ponatinib PO daily. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Blinatumomab; Drug: Cytarabine; Drug: Methotrexate; Drug: Ponatinib

INTERVENTIONS:
Biological: Blinatumomab — Given IV
  Other Names: Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI-538; MT-103
Drug: Cytarabine — Given intrathecally via spinal tap
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Methotrexate — Given intrathecally via spinal tap
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Ponatinib — Given PO
  Other Names: AP-24534; AP24534

SUMMARY:
This phase II trial studies how well blinatumomab, methotrexate, cytarabine, and ponatinib work in treating patients with Philadelphia chromosome (Ph)-positive, or BCR-ABL positive, or acute lymphoblastic leukemia that has come back or does not respond to treatment. Immunotherapy with monoclonal antibodies, such as blinatumomab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as methotrexate and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Ponatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving blinatumomab, methotrexate, cytarabine, and ponatinib may work better in treating patients with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the complete molecular response rate in cohort 1 (newly diagnosed Philadelphia chromosome [Ph-positive] and/or BCR-ABL-positive acute lymphoblastic leukemia [ALL]) and the overall response (complete remission [CR]+CR with incomplete blood count recovery [CRi]) rate in cohort 2 (relapsed/refractory disease).

SECONDARY OBJECTIVES:

I. To evaluate other clinical efficacy endpoints (complete cytogenetic response, complete molecular response [CMR], event-free survival [EFS] and overall survival [OS]) and safety of the regimen.

EXPLORATORY OBJECTIVES:

I. To characterize the role of ABL1 kinase domain mutations on treatment failure and relapse in patients with Ph+ ALL treated with blinatumomab ponatinib.

II. To determine the impact of recurrent genomic alterations at diagnosis on relapse-free survival (RFS) in patients with Ph+ ALL treated with blinatumomab plus ponatinib.

III. To investigate the impact of next-generation sequencing-based minimal residual disease assessment on relapse-free survival in patients with Ph+ ALL.

IV. To determine the effect on immune cell subsets in patients with Ph+ ALL treated with blinatumomab plus ponatinib.

OUTLINE:

Patients receive blinatumomab intravenously (IV) nonstop on days 1-28 of cycles 1-5, and methotrexate and cytarabine intrathecally (by spinal tap) on days 1, 15, and 29 of cycles 1-4. Patients also receive ponatinib orally (PO) daily. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of one of the following:

   1. Participants ≥ 18 years of age with previously untreated Ph-positive ALL [either t(9;22) and/or BCR-ABL positive] (includes patients initiated on first course of therapy before cytogenetics known) or with lymphoid accelerated or blast phase CML. These participants could have received one or two courses of chemotherapy with or without other TKIs and still eligible. (Participants with lymphoid accelerated or blast phase CML will be evaluated separately) i. If they achieved CR, they are assessable only for event-free and overall survival, or ii. If they failed to achieve CR, they are assessable for CR, event-free, and overall survival
   2. Participants ≥ 18 years of age with relapsed/refractory Ph-positive ALL or with previously treated lymphoid accelerated or blast phase CML (Participants with lymphoid accelerated or blast phase CML will be evaluated separately)
   3. Participants ≥ 18 years of age with ALL MRD positive (either by NGS or PCR or flowcytometry) or with previously treated lymphoid accelerated or blast phase CML (Participants with lymphoid accelerated or blast phase CML will be evaluated separately)
2. Performance status ≤ 2 (ECOG Scale)
3. Adequate liver function as defined by the following criteria (unless the increased values are judged to be leukemia disease related):

   1. Total serum bilirubin ≤ 2 x upper limit of normal (ULN), unless due to Gilbert's syndrome
   2. Alanine aminotransferase (ALT) ≤ 3 x ULN, OR
   3. Aspartate aminotransferase (AST) ≤ 3 x ULN
4. Adequate pancreatic function as defined by the following criteria:

   a) Serum lipase and amylase ≤ 1.5 x ULN
5. For females of childbearing potential, a negative urine pregnancy test must be documented
6. Female participants who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse
7. Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:

   * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or
   * Agree to completely abstain from heterosexual intercourse
8. Adequate cardiac function as assessed clinically by history and physical examination.
9. Signed informed consent

Exclusion Criteria:

1. Active serious infection not controlled by oral or intravenous antibiotics.
2. History of acute pancreatitis within 1 year of study or history of chronic pancreatitis
3. History of alcohol abuse
4. Uncontrolled hypertriglyceridemia (triglycerides > 650mg/L)
5. Active secondary malignancy other than skin cancer (e.g., basal cell carcinoma or squamous cell carcinoma) that in the investigator's opinion will shorten survival to less than 1 year.
6. Active Grade III-V cardiac failure as defined by the New York Heart Association Criteria.
7. Uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

   * Myocardial infarction (MI), stroke, or revascularization within 3 months
   * Unstable angina or transient ischemic attack
   * Congestive heart failure prior to enrollment, or left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards prior to enrollment
   * Diagnosed or suspected congenital long QT syndrome
   * Clinically significant atrial or ventricular arrhythmias (such as artrial fibrillation, ventricular tachycardia, ventricular fibrillation, or Torsades de pointes) as determined by the treating physician
   * Prolonged QTc interval on pre-entry electrocardiogram (> 470 msec) unless corrected after electrolyte replacement or approved by cardiologist
   * Significant venous or arterial thromboembolism including deep venous thrombosis or pulmonary embolism. Participants with a history of treated prior superficial or catheter associated will not be considered as significant embolism and after discussion with PI will not be excluded from eligibility.
   * Uncontrolled hypertension (diastolic blood pressure >90mmHg; systolic >140mmHg). Participants with hypertension should be under treatment on study entry to effect blood pressure control
8. History or presence of clinically relevant CNS pathology or event such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis or severe (grade 3 or above) CNS events including ICANS from prior CART or other T cell engager therapies. Participants with active CNS leukemia - will NOT be excluded
9. Current autoimmune disease or history of autoimmune disease with potential CNS involvement
10. Treatment with any investigational antileukemic agents or chemotherapy agents within 2 weeks prior to study entry, unless full recovery from side effects has occurred or participant has rapidly progressive disease judged to be life-threatening by the investigator.
11. Pregnant and lactating women will not be eligible; women of childbearing potential should have a negative pregnancy test prior to entering on the study and be willing to practice methods of contraception. Women do not have childbearing potential if they have had a hysterectomy or are postmenopausal without menses for 12 months. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control.
12. History of significant bleeding disorder unrelated to cancer, including:

    * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
    * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
13. Participants with documented significant pleural or pericardial effusions unless they are thought to be secondary to their leukemia.
14. Known active infection with HIV, HBV, HCV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Complete molecular response (CMR) rate in newly diagnosed Ph-positive and/or BCR-ABL-positive acute lymphoblastic leukemia (ALL) | At 18 weeks
Overall response rate (ORR) in relapsed/refractory ALL | At 12 weeks
  This is defined as the percentage of patients achieving complete remission (CR) or CR with incomplete blood count recovery (CRi).
Relapse-free survival | From documented complete response until relapse or death, assessed up to 6 years
Event-free survival | From first day of treatment until any failure (resistant disease, relapse, or death), assessed up to 6 years
Overall survival | First day of treatment to time of death from any cause, assessed up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Short NJ, Kantarjian H, Furudate K, Jain N, Ravandi F, Karrar O, Loghavi S, Nasr L, Haddad FG, Senapati J, Garris R, Takahashi K, Jabbour E. Molecular characterization and predictors of relapse in patients with Ph + ALL after frontline ponatinib and blinatumomab. J Hematol Oncol. 2025 May 14;18(1):55. doi: 10.1186/s13045-025-01709-y. PMID 40369607
- [Derived] Kantarjian H, Short NJ, Haddad FG, Jain N, Huang X, Montalban-Bravo G, Kanagal-Shamanna R, Kadia TM, Daver N, Chien K, Alvarado Y, Garcia-Manero G, Issa GC, Garris R, Nasnas C, Nasr L, Ravandi F, Jabbour E. Results of the Simultaneous Combination of Ponatinib and Blinatumomab in Philadelphia Chromosome-Positive ALL. J Clin Oncol. 2024 Dec 20;42(36):4246-4251. doi: 10.1200/JCO.24.00272. Epub 2024 Jul 19. PMID 39028925
- [Derived] Jabbour E, Short NJ, Jain N, Huang X, Montalban-Bravo G, Banerjee P, Rezvani K, Jiang X, Kim KH, Kanagal-Shamanna R, Khoury JD, Patel K, Kadia TM, Daver N, Chien K, Alvarado Y, Garcia-Manero G, Issa GC, Haddad FG, Kwari M, Thankachan J, Delumpa R, Macaron W, Garris R, Konopleva M, Ravandi F, Kantarjian H. Ponatinib and blinatumomab for Philadelphia chromosome-positive acute lymphoblastic leukaemia: a US, single-centre, single-arm, phase 2 trial. Lancet Haematol. 2023 Jan;10(1):e24-e34. doi: 10.1016/S2352-3026(22)00319-2. Epub 2022 Nov 16. PMID 36402146
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org